CLINICAL TRIAL: NCT06737874
Title: Predictive Value of Revised Trauma Score(RTS)and Glasgow Coma Scale (GCS)of Mortality in Patients with Multiple Trauma in Emergency Department At Assiut University Hospital & Ismailia University Hospitals.
Brief Title: Predictive Value of Revised Trauma Score(RTS)and Glasgow Coma Scale (GCS)of Mortality in Patients with Multiple Trauma.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abd Elrhman Salah Abuozied Mansour, Doctor, Assiut University
Other Study IDs: RTS & GCS in trauma patients
Record Dates: First submitted 2024-12-02; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Polytrauma Patients
Keywords: Predictive value of Revised Trauma Score(RTS)and Glasgow Coma Scale (GCS)of mortality in patients with multiple trauma in emergency department

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group A: polytrauma patients

SUMMARY:
This study aims to assess the efficacy of RTS and GCS in predicating the mortality among multiple trauma patients admitted to emergency departments at Assiut university hospital.Which score is better in predicting mortality in polytrauma patients Revised Trauma Score (RTS) or Glasgow Coma Scale (GCS) of with Multiple Trauma?

DETAILED DESCRIPTION:
Trauma is a serious global health problem. Globally around 5.8 million people deaths were estimated from injuries in 2004. These deaths accounted for 10% of the world's mortality[1]. It is the fifth leading cause ofsignificant, disability and sixth leading cause of death[2]. More than 90% of the world's injury deaths occur in low- and middle-income countries[3]. Injury deaths in Egypt accounted for 8% and the eighth leading cause of death in 2010[4]. There was an increase in the number of hospitalization due to trauma. In Upper Egypt, trauma cases increased from 19,869 up to 32,699 with death rate 1.2/100 cases per year throughout the period from 2002 to 2009.In multiple trauma patient management, time is crucial. Early intervention has consistently been shown to reduce mortality and morbidity[5]. Prompt and effective care [6]. These scores either measure the alteration in patient's physiology; Glasgow Coma Scale (GCS) and Revised Trauma Score (RTS) or anatomy; Injury Severity Score (ISS)[7]. Glasgow Coma Scale (GCS) is one of the most commonly used trauma scores and is a good predictor of the outcome. The GCS is primarily utilized to evaluate the level of consciousness impairment in patients, achieved through the assessment of ocular, motor, and verbal response[8].The Revised Trauma Score (RTS) are considered the most practical and effective [9].The RTS stands out because it can be quickly calculated using a patient's initial clinical status and vital signs at presentation, making it particularly useful during the critical "golden hour" after arrival[10]

ELIGIBILITY:
Inclusion Criteria:

* 1-patients aged from > 18 years old. 2-Both male and female. 3-Patients have penetrating and blunt trauma.

Exclusion Criteria:

* 1-Pregnant women. 2-Patients with mild trauma such as soft tissue damage and 3-isolated limb fractures. 4-Patients were transferred to another hospital. 5-Failure of follow-up for any reason. 6-Patients who refused participatioc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multiple trauma patients admitted to Emergency department. The Berlin definition defines polytrauma as a life-threatening injury involving at least 2 bodily regions (each with an AIS ≥3) as well as at least one positive physiologic parameter. The physiologic parameters include the elderly (age ≥70 years), low systolic blood pressure, Glasgow coma score ≤8, coagulopathy, and acidosis[17].
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 30 day
  to identify the trauma-related mortality rate among patients

SECONDARY OUTCOMES:
Admission | 30days
  Associated risk factors that affect multiple trauma patient's outcome. Outcome of patients :(death/survival) with 30 day of admission , hospital stay, and ICU admission